CLINICAL TRIAL: NCT06693245
Title: Observation of Pain During the Treatment of Great Saphenous Vein Using Microwave Ablation， and Analysis of Related Factors
Status: Recruiting | Type: Observational
Sponsor: Chengdu University of Traditional Chinese Medicine (Other)
Responsible Party: Principal Investigator, Chunshui He, chief physician, Chengdu University of Traditional Chinese Medicine
Other Study IDs: ChengduUTCMvs7
Record Dates: First submitted 2024-11-14; First posted 2024-11-18 (Actual); Last update posted 2024-11-18 (Actual); Status verified 2024-11

CONDITIONS: Vascular Disease，Peripheral; Venous Insufficiency of Leg; Varicose Veins of Lower Limb
Keywords: Varicose veins of the lower extremities; Endovenous Microwave Ablation; intraoperative pain; visual analogue scale of pain
MeSH Terms: conditions — Peripheral Vascular Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Observation of Pain and Analysis of Related Factors During Microwave Ablation Treatment of Saphenous: Among 155 patients, our team measured the diameter of the great saphenous vein preoperatively according to the CEAP classification and ultrasound measurements. We performed endovenous microwave ablation of the great saphenous vein along with foam sclerotherapy and point stripping treatment. We documented the operating room temperature, puncture site, VAS scores during puncture and catheter placement, the amount of injected tumescent fluid, radiofrequency generator used, and data at the conclusion of the surgery. A descriptive analysis of intraoperative pain scores was conducted to evaluate the level of pain experienced during the surgery. A nonparametric test was utilized to analyze the relationship between preoperative and intraoperative factors and the level of pain experienced during the surgery.
  Interventions: Procedure: VAS scores of the puncture

INTERVENTIONS:
Procedure: VAS scores of the puncture — All patients were evaluated by our team with CEAP grading and ultrasound measurements to record the diameter of the saphenous vein before surgery。We performed endovenous microwave ablation of the great saphenous vein along with foam sclerotherapy and point stripping treatment. We documented the operating room temperature, puncture site, VAS scores during puncture and catheter placement, the amount of injected tumescent fluid, radiofrequency generator used, and data at the conclusion of the surgery. A descriptive analysis of intraoperative pain scores was conducted to evaluate the level of pain experienced during the surgery. A nonparametric test was utilized to analyze the relationship between preoperative and intraoperative factors and the level of pain experienced during the surgery.

SUMMARY:
Objective: This study is a single-center prospective observational research that recorded patients' pain scores at four time points during surgery (puncture and catheter insertion, swelling fluid injection, microwave generator operation, and end of surgery). It analyzed the correlation between pain during microwave ablation treatment for great saphenous vein varicosities and factors such as age, gender, body mass index, volume of swelling fluid used, and others, in order to summarize and improve surgical details to reduce patients' intraoperative pain.

DETAILED DESCRIPTION:
Despite the significant progress made by global experts in vascular surgery in studying endovenous microwave ablation (EMA) for the treatment of varicose veins (VVs), there are still many unknown areas to be explored. Current research primarily focuses on the surgical outcomes and associated complications of EMA, while studies on intraoperative pain are relatively scarce. Firstly, the American College of Radiology has not provided a clear definition of intraoperative pain when treating lower extremity varicose veins, thus it has not received sufficient attention in clinical practice. Many physicians consider the success of the surgery as the endpoint of treatment, overlooking the impact of intraoperative pain on the patient's surgical experience. Ni Zhao et al. found in a prospective randomized controlled trial that EMA is associated with more pain within 48 hours post-operation. When our department introduced the use of EMA for VVs, we discovered that its working form and power differ from other thermal ablations, and there are also differences in terms of intraoperative pain, the volume of tumescent fluid used, and the requirements for vein depth. With the continuous advancement in lower limb varicose vein surgeries, anesthesia methods have evolved from general anesthesia to combined spinal-epidural anesthesia, and now to local anesthesia. Tumescent anesthetic solution is the main anesthetic agent for EMA surgery, and the infiltration of tumescent anesthetic fluid around the great saphenous vein is crucial for the success of EMA; however, paradoxically, this is also the area where patients experience the most severe pain. The commonly used tumescent solution is a crystalline solution containing local anesthetics and adrenaline, which is acidic in nature and is the main reason for the 'sting' sensation during skin infiltration. A Cochrane review indicated that adjusting the pH of lidocaine solution by adding sodium bicarbonate significantly reduced pain during the skin infiltration process, as measured by the 10-centimeter Visual Analog Scale (VAS). Moreover, the temperature of the tumescent anesthetic solution also affects pain during the skin infiltration process, as noted by Bell et al. Alonso et al. found in a prospective randomized controlled trial that heating local anesthetic solutions to 37°C and 42°C can reduce pain, and heating adrenaline-containing local anesthetic solutions to near body temperature is also an effective method to alleviate local anesthetic pain. We hope to achieve better preoperative prevention and intraoperative management through an analysis of pain-related factors, thereby improving the patient's surgical experience.

ELIGIBILITY:
Inclusion Criteria:

1. Age≥ 18 years old, ≤ 90 years old;
2. the patient's life expectancy is greater than 12 months;
3. The clinical diagnosis is primary VVs, CEAP classification C2-C6, and the GSV segment needs to be treated, including pain, burning sensation, heaviness, fatigue, itchy skin, night cramps and other clinical symptoms;
4. Doppler ultrasound confirmed that the diameter of GSV was greater than 3mm and less than 12mm when standing;
5. Doppler ultrasound confirms that GSV is located in the saphenofascia or the distance between GSV and the skin surface is >1cm;
6. endovenous microwave ablation treatment only for unilateral GSV walking area;
7. The patient is willing to cooperate with the completion of the examination specified in the protocol.

Exclusion Criteria:

1. GSV thrombosis, or combined with deep vein thrombosis, or previous history of deep vein thrombosis and pulmonary embolism;
2. patients with recurrence after prior VVs-related surgery (C2r);
3. the GSV trunk is severely distorted, and it is expected that the catheter will not be able to pass;
4. Severe ischemia of the lower limbs, Ankle brachial pressure index (ABPI) < 0.8;
5. Known allergy to the drugs and device materials involved in the study;
6. Previously implanted with a pacemaker or defibrillator, and currently receiving regular anticoagulation therapy (such as warfarin, heparin);
7. Pregnant or lactating females;
8. Patients who are unable or unwilling to participate in the study;
9. Participating in the research of other drugs or devices;
10. Skin malignancies other than non-melanoma that are being treated;
11. daily use of narcotic drugs or non-steroidal anti-inflammatory drugs to control pain caused by venous disease;
12. The investigator judged that endovenous treatment was not suitable;

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with primary VVs from December 2024 to December 2025 who were admitted to the hospital and underwent endovenous microwave ablation treatment for the main trunk of the saphenous vein
Sampling Method: Probability Sample
Enrollment: 155 (Estimated)
Dates: Start 2024-12-01 (Estimated); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Visual Analogue Scale (VAS) Pain Score | during operation
  We mainly record the VAS pain scores during local anesthetic injection, needle puncture, catheter placement, swollen anesthetic injection, microwave generator operation, and at the end of the surgery.
Basic data related to surgery | intraoperative
  We also documented the patient's heart rate, blood pressure, oxygen saturation, along with the temperature of the operating room, location of puncture, number of incisions, and volume of injected swelling fluid, among others. These data are recorded to explore their correlation with the intraoperative VAS pain score.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital of Chengdu University of Traditional Chinese Medicine, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yang X, Li J, Bai X, Zhou L, Xu W. Endovenous Microwave Ablation Versus Radiofrequency Ablation for the Treatment of Lower Limb Varicose Veins. Ann Vasc Surg. 2024 Jan;98:301-308. doi: 10.1016/j.avsg.2023.06.024. Epub 2023 Jul 7. PMID 37423329
- [Background] Nandhra S, Wallace T, El-Sheikha J, Leung C, Carradice D, Chetter I. A Randomised Clinical Trial of Buffered Tumescent Local Anaesthesia During Endothermal Ablation for Superficial Venous Incompetence. Eur J Vasc Endovasc Surg. 2018 Nov;56(5):699-708. doi: 10.1016/j.ejvs.2018.05.017. Epub 2018 Jun 29. PMID 30392525
- [Background] Usach I, Martinez R, Festini T, Peris JE. Subcutaneous Injection of Drugs: Literature Review of Factors Influencing Pain Sensation at the Injection Site. Adv Ther. 2019 Nov;36(11):2986-2996. doi: 10.1007/s12325-019-01101-6. Epub 2019 Oct 5. PMID 31587143
- [Background] Cepeda MS, Tzortzopoulou A, Thackrey M, Hudcova J, Arora Gandhi P, Schumann R. Adjusting the pH of lidocaine for reducing pain on injection. Cochrane Database Syst Rev. 2010 Dec 8;(12):CD006581. doi: 10.1002/14651858.CD006581.pub2. PMID 21154371
- [Background] Anuforo A, Evbayekha E, Agwuegbo C, Okafor TL, Antia A, Adabale O, Ugoala OS, Okorare O, Phagoora J, Alagbo HO, Shamaki GR, Disreal Bob-Manuel T. Superficial Venous Disease-An Updated Review. Ann Vasc Surg. 2024 Aug;105:106-124. doi: 10.1016/j.avsg.2024.01.009. Epub 2024 Apr 5. PMID 38583765
- [Background] Li Y, Wu W, Li Y, Li J, Sun M. Efficacy and safety of endovenous microwave ablation versus laser ablation for great saphenous vein varicosis: study protocol for a multicentre, randomised controlled non-inferiority trial. BMJ Open. 2022 May 25;12(5):e059213. doi: 10.1136/bmjopen-2021-059213. PMID 35613801
- [Background] Hu J, Zhao T, Geng W, Lu Y, Zhao XF, Li YZ, Tang YQ, Liu JW, Wang LY, Janiak C, Yang XY, Su BL. Correction: Synthesis of hydrophobic and hydrophilic TiO2 nanofluids for transformable surface wettability and photoactive coating. Chem Commun (Camb). 2019 Sep 24;55(77):11642. doi: 10.1039/c9cc90390a. PMID 31512684